CLINICAL TRIAL: NCT01540695
Title: Does Cryofixation of Skin Specimens Affect Quality of Subsequent Formalin Fixed Paraffin Embedded H&E Histology
Brief Title: Does Cryofixation of Skin Specimens Affect Quality of Subsequent Formalin Fixed Paraffin Embedded H and E Histology
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 25911
Record Dates: First submitted 2012-02-09; First posted 2012-02-29 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Basal Cell Carcinoma; Squamous Cell Carcinoma
Keywords: Any patient with a routine basal cell or squamous cell carcinoma; of the skin diagnosed on frozen histology during a Mohs procedure
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This prospective study of 60 slides of basal and squamous cell carcinomas of the skin aims to determine whether:

1. The process of cryofixation prior to generating formalin fixed paraffin embedded (FFPE) H&E sections alters the histology in skin tumor specimens.
2. Which specific histologic parameters are altered between previously cryofixed versus routine FFPE sections. Histologic observations will be recorded by two dermatopathologists and two Mohs surgeons and statistically analyzed.

DETAILED DESCRIPTION:
Generating formalin fixed paraffin embedded (FFPE) hematoxylin and eosin (H&E) stained permanent sections from previously cryofixed tissue is a common practice used to confirm diagnosis of frozen section histology. In dermatology, this practice can be used to examine Mohs layers and its debulk as well as routine nonmelanoma skin cancer (NMSC) biopsies after initial histologic diagnosis with frozen sections. Even though freezing tissue can introduce histologic artifacts, there have been no studies documenting whether this occurs specifically in cryofixed tissues that are subsequently thawed for permanent FFPE H&E histology. The purpose of our study is to determine whether the freeze-thaw process used to generate permanent sections after cryofixation introduces significantly detectable histologic differences compared to permanent sections that were not previously cryofixed. Thirty debulk specimens of basal cell and squamous cell carcinomas will be prospectively collected. Each specimen will be split so that half is processed as cryofixed permanents and the other half as noncryofixed permanents. The investigator will show each slide in random order to a group of four blinded participants (two dermatopathologists and two Mohs surgeons). Each participant must first rate the overall quality of histology. Then, each participant will rate each slide on the quality of cellular morphology, nuclear morphology, color and contrast of stains, intactness of specimen, and other miscellaneous artifacts. These data will then be analyzed for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18 or over) with a biopsy proven routine basal cell or squamous cell carcinoma of the skin who are scheduled for treatment with the Mohs procedure by Dr. Christopher Miller at the University of Pennsylvania's Division of Dermatologic Surgery will be included. Both female and male patients will be included.

Exclusion Criteria:

* Patients with basal cell or squamous cell carcinomas of more complex histopathology will be excluded from the study. Complex histopathology of a tumor is defined as features with aggressive, moderately to poorly differentiated, or unusual histopathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients will be recruited from the Mohs unit of the HUP Department of Dermatology
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2012-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | October 2016 to March 2018

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Miller, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramsonc Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States